CLINICAL TRIAL: NCT03723681
Title: A Study to Evaluate the Safety and Pharmacokinetics of Quizartinib in Combination With Standard Induction Therapy and Consolidation Therapy in Chinese Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Study of Quizartinib in Combination With Standard Therapies in Chinese Participants With Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-A103
Record Dates: First submitted 2018-10-18; First posted 2018-10-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quizartinib 20 mg (Experimental): Participants receive 20 mg quizartinib in combination with standard induction therapy and consolidation therapy once daily in the fasted state in the morning (at least 1 hour before or two hours after a meal)
  Interventions: Drug: Quizartinib
- Quizartinib 40 mg (Experimental): Participants receive 40 mg quizartinib in combination with standard induction therapy and consolidation therapy once daily in the fasted state in the morning (at least 1 hour before or two hours after a meal)
  Interventions: Drug: Quizartinib

INTERVENTIONS:
Drug: Quizartinib — Quizartinib is provided as 20 mg tablets for oral administration
  Other Names: Experimental product; AC220

SUMMARY:
20 mg or 40 mg of quizartinib will be given to Chinese patients who were just diagnosed with AML. The study drug will be given to them along with standard therapies. The purpose is to find out the highest dose they can stand.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label study to evaluate the safety and pharmacokinetics (PK) of quizartinib in combination with standard induction therapy and consolidation therapy in Chinese patients with newly diagnosed AML.

The quizartinib doses will be Level 1: 20 mg and Level 2: 40 mg. No increase in the quizartinib dose will be made in the same subject.

Dose-limiting toxicity associated with quizartinib occurring at each level will be assessed, and the maximum tolerated dose (MTD) will be decided using a 3 + 3 design.

ELIGIBILITY:
Inclusion criteria:

* Has provided written informed consent for participation in the study
* Is aged 18 to 70 years at the time of enrollment into the study
* Has newly diagnosed, morphologically documented primary AML or AML secondary to myelodysplastic syndrome or a myeloproliferative neoplasm based on the World Health Organization (WHO) 2008 classification (at Screening)
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 at enrollment
* Has all of the required laboratory test results performed within 14 days prior to enrollment in the study.
* Is capable of orally taking quizartinib
* Is capable of being admitted to the hospital during the dose limiting toxicity (DLT) evaluation period
* If a woman of childbearing potential, has a negative serum pregnancy test upon entry into this study and is willing to use highly effective birth control upon enrollment, during the treatment period and for 6 months following the last dose of investigational drug or cytarabine, whichever is later. A woman is considered of childbearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (having undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy).
* If male, is surgically sterile or willing to use highly effective birth control upon enrollment, during the treatment period, and for 6 months following the last dose of investigational drug or cytarabine, whichever is later.

Exclusion criteria:

* Has diagnosis of acute promyelocytic leukemia (APL), French-American-British classification M3 or WHO classification of APL with translocation, t(15;17)(q22;q12), or BCR-ABL positive leukemia (ie, chronic myelogenous leukemia in blast crisis). Subjects who undergo diagnostic workup for APL and treatment with all-trans retinoic acid (ATRA), but who are found not to have APL, are eligible (treatment with ATRA must be discontinued before starting induction chemotherapy).
* Has a diagnosis of AML secondary to prior chemotherapy or radiotherapy for other neoplasms
* Had prior treatment for AML, except for the following allowances:

  1. Leukapheresis
  2. Treatment for hyperleukocytosis with hydroxyurea
  3. Cranial radiotherapy for central nervous system (CNS) leukostasis
  4. Prophylactic intrathecal chemotherapy
  5. Growth factor or cytokine support
* Has received prior treatment with any investigational product or device within 30 days prior to enrollment in the study or is currently participating in other investigational procedures
* Has a history of other malignancies excluding the following:

  1. Adequately treated non-melanoma skin cancer
  2. Curatively treated in situ disease, or other solid tumors curatively treated with no evidence of disease for at least two years
* Has a past or current history of the following cardiovascular diseases:

  1. Heart rate of < 50 beats/min performed with 12-lead ECG within 14 days prior to enrollment in the study (excluding patients using a heart pacemaker)
  2. QT interval corrected by Fridericia (QTcF) of ≥ 450 msec performed with 12-lead ECG within 14 days prior to enrollment in the study
  3. Congenital long QT syndrome diagnosed or suspected (including family history of long QT syndrome)
  4. Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg measured within 7 days prior to enrollment in the study
  5. History of clinically significant ventricular arrhythmias [such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes (TdP)]
  6. History of second (Mobitz II) or third-degree heart block (patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker)
  7. History of uncontrolled angina pectoris or myocardial infarction within 6 months prior to enrollment in the study
  8. History of heart failure according to New York Heart Association (NYHA) Functional Classification: Class 3 or 4 heart failure
  9. Left ventricular ejection fraction (LVEF) of ≤ 45% or lower than the institutional lower limit of normal value per multi-gated acquisition scan (MUGA) or echocardiogram done within 30 days prior to enrollment
  10. Complete left bundle branch block
* Has active acute or chronic systemic fungal, bacterial, or viral infection not well controlled by antifungal, antibacterial, or antiviral therapy
* Has active clinically relevant liver disease (such as active hepatitis B or active hepatitis C).
* Has a history of human immunodeficiency virus (HIV). Patients will be tested for HIV prior to enrollment in the study, if required by local regulations or the Ethics Committee.
* Has a history of hypersensitivity to any excipients in the quizartinib tablets
* Is a female who is pregnant or breastfeeding
* Is considered inappropriate for the study by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities | At the end of induction phase at approximately 56 days
Number of Participants with Adverse Events During the Trial | within approximately 19 months
Maximum Concentration (Cmax) | within 56 days
  Categories: quizartinib, active metabolite
Time to Cmax (Tmax) | within 56 days
  Categories: quizartinib, active metabolite
Area under the Plasma Concentration-Time Curve (AUC) | within 56 days
  Categories: quizartinib, active metabolite

SECONDARY OUTCOMES:
Number of Participants with Response | within approximately 19 months
  Categories: Complete remission (CR), CR with incomplete platelet or hematological recovery (CRi), partial remission (PR), no response (NR)
Response Rates | within approximately 19 months
  Categories: response rate (CRc + PR), composite CR (CRc: CR + CRi) rate

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/